CLINICAL TRIAL: NCT05759247
Title: Evaluation of the Use of a Remote Monitoring and Follow-up Option for Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Evaluation of the Use of a Remote Monitoring and Follow-up Option for Patients With Chronic Obstructive Pulmonary Disease (BOREAL)
Acronym: BOREAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Biosency (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP211098; 2021-A02146-35 (Other: ID-RCB Number)
Record Dates: First submitted 2023-01-19; First posted 2023-03-08 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; acute exacerbation; prevention; early detection
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BORA Band (wristband) — Wristband collecting patient vital signs and activity

SUMMARY:
The purpose of this study is to evaluate the ability of the Bora Care remote monitoring solution to detect early acute exacerbations of Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Worldwide, COPD has been increasing for 20 years with nearly 300 million patients, i.e. 4 to 10% of the adult population (7.5% in France). According to the WHO, it is now the fourth leading cause of death in the world.

Acute exacerbations of COPD (worsening of symptoms requiring an increase in treatment) represent frequent events in the course of the disease and the consequences are significant for the patient in terms of vital prognosis, deterioration of respiratory function, impact on quality life and for the health system in terms of cost. Missed diagnosis and delayed treatment are associated with impaired outcomes. The prevention and early treatment of acute exacerbations of COPD therefore have a major role in the management of COPD patients and could be facilitated by telemonitoring tools.

The purpose of the present study is to validate the interest of remote monitoring of various parameters (cardio-respiratory, environmental, symptom questionnaires) to predict and detect early the occurrence of acute exacerbations of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patient with COPD defined according to the SPLF recommendations, whose level of lung function in a stable state is known (measurement less than 12 months old)
* Patient with at least one of the following criteria :

  * Hospitalized for a COPD exacerbation at the time of enrolment in the study, and having had at least one other exacerbation in the last 12 months
  * Followed-up and part of the active file of the site, having had at least 2 exacerbations during the last 12 months, including one with hospitalization
  * COPD patient with at least 2 exacerbations in the last 12 months, including one with hospitalization
* Patient having given written informed consent to participate in the study
* Patient affiliated to the French social security system

Exclusion Criteria

* Vulnerable patient (minor, protected adult, prisoner)
* Patient unable to use the BoraBand tool and without access to a caregiver
* Presence of a comorbidity considered unstable or very severe by the investigator
* Patient already participating in another interventional research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Performance of the device for early detection of AECOPD | 12 months
  Sensibility and specificity of the alerts computed for all AECOPD event recorded in the study

SECONDARY OUTCOMES:
Relation between AECOPD and measured parameters | 12 months
  Correlation between measured parameters and observed AECOPD events
Compliance | 12 months
  Wristband wearing duration during the follow-up period
Description of AECOPD | 12 months
  Number, duration, severity of AECOPD events observed during the study
Quality of Life CAT | 12 months
  Quality of life questionnaire CAT at baseline and after 6 and 12 months - CAT : COPD Assement Test, 8 items, range 0 (no impact of COPD) - 40 (worst impact of COPD)
Quality of Life EQ5D5L | 12 months
  Quality of life questionnaire EQ5D5L at baseline and after 6 and 12 months - EQ5S5L : five dimensions, 5 levels each, final result expressed as a 5-digit number that describes the patient's health state (worsens with increasing score)
Satisfaction | 12 months
  meCUE questionnaire after 12 months
Symptoms - EXASCORE questionnaire | 12 months
  EXASCORE questionnaire at baseline and after 6 and 12 months. EXASCORE: 2 dimensions, 8 items, range 0-32 (the highest the worst)
Symptoms - EXACT E-RS questionnaire | 12 months
  EXACT E-RS questionnaire at baseline and after 6 and 12 months. EXACT E-RS : 4 sections, 14 items, range 0-100 (the highest the worst)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pneumology Department - Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No